CLINICAL TRIAL: NCT01425164
Title: Ischemia In Hemodialysed Patients And Outcome: Ivabradine Versus Carvedilol. A Randomized, Double Blind Study
Brief Title: Ischemia In Hemodialysed Patients: Ivabradine Versus Carvedilol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Gennaro Cice, Responsible Cardiology Unit ℅ Cappella Cangiani, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IVA-ISCHEMIA
Record Dates: First submitted 2011-08-10; First posted 2011-08-29 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Heart Disease; Angina; Hemodialysis
Keywords: hemodialysis; coronary heart disease; angina; betablocker; carvedilol; ivabradine
MeSH Terms: conditions — Coronary Disease; Angina Pectoris | interventions — Ivabradine; Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Active Comparator)
  Interventions: Drug: Carvedilol
- Ivabradine (Experimental)
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — ivabradine tablets, 5 to 7.5 mg bis-in-die.
  Arms: Ivabradine
Drug: Carvedilol — carvedilol tablets, 12.5 to 25 mg bis-in-die.
  Arms: Carvedilol

SUMMARY:
In hemodialysed patients, coronary heart disease is the leading cause of mortality and morbidity. Most of the commonly used drug for ischemia are used in this patients, but few prospective data are available. Among anti-ischemic drugs betablocker provided evidence of beneficial effects on outcome and, in dialysis patients, carvedilol was successfully used also in heart failure. Ivabradine is the latest anti-ischemic drug that provided evidence of benefit in general population, but no study is available in dialysis patients. Aim of the present study is to compare in a randomized, double-blind, parallel group trial the effects of ivabradine compared with carvedilol on event-free survival at 18 months in a hemodialysed population of patients with established coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* documented CAD evidenced by either coronary angiography (>50% diameter stenosis of a major coronary artery) or a previously documented myocardial infarction
* transient ischemia evidenced by abnormalities during an exercise ECG (standard Bruce protocol), myocardial perfusion scintigraphy, or stress regional wall motion study done within 6 months of study entry

Exclusion Criteria:

* unstable angina pectoris
* myocardial infarction or coronary revascularization within 3 months of study entry
* an ECG abnormality interfering with exercise ST-segment interpretation (eg, ST-segment depression >0.5 mm, QRS duration >0.1 second, R-wave amplitude <8 mm,preexcitation,or atrial fibrillation)
* inability to undergo exercise testing
* uncontrolled hypertension
* other serious condition (medical, psychiatric, cognitive, or social)
* symptoms of sufficient severity (Canadian class II or higher) to require antianginal medications other than nitrates
* heart failure
* greater than first-degree atrio-ventricular block, asthma, or other contraindications to betablocker therapy

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
event-free survival | 18 months
  primary outcome was event-free survival at 18 months. The following ischemia related events were considered: death, resuscitation from ventricular tachycardia/fibrillation, nonfatal myocardial infarction, hospitalization for unstable angina, aggravation of angina requiring known antianginal therapy, and need for revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Cice, MD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Chair of Cardiology Second University of Naples, Naples, Italy